CLINICAL TRIAL: NCT06134505
Title: Evaluation of the Efficiency of Local Application of Bee Products in the Care of Diaper Dermatitis in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, İlknur KAHRİMAN, Assoc. Prof, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: İlknurKahriman
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Diaper Dermatitis Healing
Keywords: diaper dermatitis; healing; bee products; care
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Experimental Group1 (Experimental): Barrier cream group 1 consists of a mixture of propolis, beeswax, queen bee larva and plant oil
  Interventions: Procedure: Use of Barrier cream group 1 in the healing of diaper dermatitis
- Experimental: Experimental Group2 (Experimental): Olive oil group
  Interventions: Procedure: Use of olive oil in the healing of diaper dermatitis
- Control Group (Active Comparator): Barrier cream group 2 consists of zinc oxide
  Interventions: Procedure: Use of Barrier cream 2 in the healing of diaper dermatitis

INTERVENTIONS:
Procedure: Use of Barrier cream group 1 in the healing of diaper dermatitis — In this study, the infant's first-degree diaper dermatitis was determined by the doctor or midwife using the Uncomplicated Diaper Dermatitis Severity Rating Scale in Infants. After first-degree diaper dermatitis was detected in the babies and their written consent was obtained, the parents of the babies were informed about the research before application and the parent-baby identification information form was filled out. Families were provided with education based on the ABCDE model. Mothers were informed that Barrier cream 1 would be used at each diaper change. Baby dermatitis was monitored face to face by the researcher on the 1st, 3rd and 5th days, and the scores were recorded on the observation form. Follow-up of those with a diaper dermatitis score of "0" was discontinued because full recovery was achieved.
  Arms: Experimental: Experimental Group1
Procedure: Use of Barrier cream 2 in the healing of diaper dermatitis — In this study, the infant's first-degree diaper dermatitis was determined by the doctor or midwife using the Uncomplicated Diaper Dermatitis Severity Rating Scale in Infants. After first-degree diaper dermatitis was detected in the babies and their written consent was obtained, the parents of the babies were informed about the research before application and the parent-baby identification information form was filled out. Families were provided with education based on the ABCDE model. Mothers were informed that barrier cream 2 would be used at each diaper change. Baby dermatitis was monitored face to face by the researcher on the 1st, 3rd and 5th days, and the scores were recorded on the observation form. Follow-up of those with a diaper dermatitis score of "0" was discontinued because full recovery was achieved.
  Arms: Control Group
Procedure: Use of olive oil in the healing of diaper dermatitis — In this study, the infant's first-degree diaper dermatitis was determined by the doctor or midwife using the Uncomplicated Diaper Dermatitis Severity Rating Scale in Infants. After first-degree diaper dermatitis was detected in the babies and their written consent was obtained, the parents of the babies were informed about the research before application and the parent-baby identification information form was filled out. Families were provided with education based on the ABCDE model. Mothers were informed that olive oil would be used at each diaper change. Baby dermatitis was monitored face to face by the researcher on the 1st, 3rd and 5th days, and the scores were recorded on the observation form. Follow-up of those with a diaper dermatitis score of "0" was discontinued because full recovery was achieved.
  Arms: Experimental: Experimental Group2

SUMMARY:
The aim of this study was to evaluate the local application of bee products in the care of diaper dermatitis in infants.

1. H1: Barrier cream 1, consisting of a mixture of propolis, beeswax, queen bee larva and plants oil used in the care of diaper dermatitis, is more effective in recovering diaper dermatitis than barrier cream 2 containing zinc oxide.
2. H2: Barrier cream 1, consisting of a mixture of propolis, beeswax, queen bee larva and plants oil used in the care of diaper dermatitis, is more effective in recovering diaper dermatitis than olive oil.
3. H3: Diaper Dermatitis Severity Assessment Scale scores are lower in babies who use barrier cream 1, which consists of a mixture of propolis, beeswax, queen bee larva and plants oil, in the care of diaper dermatitis, compared to babies who use barrier cream 2, which contains zinc oxide.
4. H4: Diaper Dermatitis Severity Assessment Scale scores are lower in babies who use barrier cream 1, which consists of a mixture of propolis, beeswax, queen bee larva and plants oil, in the care of diaper dermatitis, than babies who use olive oil.

DETAILED DESCRIPTION:
Diaper dermatitis is one of the most common dermatological problems of infancy. Diaper dermatitis constitute from approximately 25% of visits to primary health care services for dermatological complaints in the first year of life. The ABCDE rule is based on the prevention of diaper dermatitis. According to ABCDE rule; airing the bottom of babies with diaper dermatitis, changing diapers hourly in the newborn period, every 3-4 hours in infancy, cleaning using warm water or wet wipes sucked with water, applying barrier creams in a thin layer after cleaning the area, and protecting from diaper dermatitis and providing diaper hygiene. Families should be educated on the right skin care practices. This thesis study was conducted in a randomized control experimental design in order to investigate the effect of olive oil, 40% zinc oxide, propolis, royal jelly, perga and plant oil mixture on the healing process in the care of 1-6 months old infants with first degree diaper dermatitis who applied to the Family Health Center/ Child Outpatient Clinic. The population of the study will be 1-6 month old babies with first degree diaper dermatitis who are registered to Family Health Centers in Antalya's Kumluca district and applied to the pediatric outpatient clinic of Kumluca State Hospital. The sample of the study was consisted of 93 infants (Olive oil: 31, propolis, beeswax, queen bee larva and plant oil mixture: 31, 40% zinc oxide cream: 31) registered to the Family Health Center and and applied to Kumluca State Hospital between January 2022 and December 2023, aged 1-6 months and meeting the sample selection criteria. The data were collected using the "Parent-Infant Descriptive Information Form", "Observation Forms", and "Assessing the Severity of Uncomplicated Diaper Dermatitis" in Infants Scale in Infants, after obtaining the permission of the ethics committee and institution of the research. The data was evaluated using the SPSS 23 package program.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 1-6 months registered at Family Health Centers No. 1, No. 2 and No. 3,
* Infants aged 1-6 months admitted to Kumluca State Hospital's Pediatric Outpatient Clinic,
* Infants with grade one diaper dermatitis according to the Uncomplicated Diaper Dermatitis in Infants Severity Rating Scale,
* Breastfed babies,
* Babies without antibiotics,
* Families who do not regularly use protective barrier cream/oil for diaper dermatitis care,
* Babies who have not started supplementary food,
* Babies with no other dermatologic or allergic skin conditions,
* Families who agreed to participate in the study were included.

Exclusion Criteria:

* Babies who are not registered to the Family Health Centers where the research was conducted,
* Newborns and babies older than 6 months who apply to the Pediatric Outpatient Clinic of Kumluca State Hospital,
* Babies who do not have first degree diaper dermatitis according to the Uncomplicated Diaper Dermatitis Severity Rating Scale in Infants,
* Babies fed with breast milk + formula or only formula,
* Babies using antibiotics,
* Families who regularly use protective barrier cream/oil in diaper dermatitis care,
* Babies who switch to solid food,
* Babies with dermatological or other allergic skin problems,
* Babies using antimycotic drugs (Ampotericin etc.),
* Babies who use a bladder for a long time,
* Babies with urinary incontinence due to diseases such as meningomyolocele and cerebral palsy,
* Families who did not agree to participate in the research were not included.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2022-12-24 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Scale for Assessing the Severity of Uncomplicated Diaper Dermatitis in Infants | 5 minutes
  The score to be received from each item of the scale varies between "0-6". The highest and lowest scores that can be obtained from the items are 0-3 points in the "Severity of Erythema or Irritation" item, 0-1 point in the "Extent of Diaper Dermatitis" item, 0-1 point in the "Papules and Pustules" item, and 0-1 point in the "Light Skin" item. It is between 0-1 points. Low total scores from the scale indicate that the severity of diaper dermatitis is low, and high scores indicate that the severity of diaper dermatitis is high.

CONTACTS AND LOCATIONS:
Overall Officials: Ilknur Kahriman, Assoc. Prof., Study Director — Karadeniz Technical University; Bahar Aksoy, MAster, Principal Investigator — Karadeniz Technical University
Locations (1):
- Antalya Provincial Directorate of Health, Antalya, Kumluca/Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 12 months after publication
Access Criteria: Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.